CLINICAL TRIAL: NCT01055691
Title: A Two Part, Open Label, Randomized, Phase I Bioequivalence Study Comparing the Fixed Dose Combination Dapagliflozin/Metformin IR Tablet (2.5 mg/850 mg or 5 mg/1000 mg) vs. the Free Combination of Dapagliflozin and Metformin IR Tablets, in Healthy Volunteers, in the Fed State
Brief Title: A Study Comparing the Amount of Metformin and After Taking a Combination Tablet vs. Separate Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1691C00002
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers; bioequivalence; dapagliflozin; metformin
MeSH Terms: interventions — dapagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Fixed dose combination dapagliflozin/metformin IR tablets followed by free combination of dapagliflozin tablet and metform IR tablet
  Interventions: Drug: Dapagliflozin/Metformin; Drug: Dapagliflozin; Drug: Metformin
- 2 (Experimental): Free combination of dapagliflozin tablet and metform IR tablet followed by fixed dose combination dapagliflozin/metformin IR tablets
  Interventions: Drug: Dapagliflozin/Metformin; Drug: Dapagliflozin; Drug: Metformin
- 3 (Experimental): Fixed dose combination dapagliflozin/metformin IR tablets followed by free combination of dapagliflozin tablet and metform IR tablet
  Interventions: Drug: Dapagliflozin/Metformin; Drug: Dapagliflozin; Drug: Metformin
- 4 (Experimental): Free combination of dapagliflozin tablet and metform IR tablet followed by fixed dose combination dapagliflozin/metformin IR tablets
  Interventions: Drug: Dapagliflozin/Metformin; Drug: Dapagliflozin; Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin/Metformin — Fixed dose combination dapagliflozin/metformin IR tablet 2.5 mg/850 mg Oral Single dose
  Arms: 1; 2
Drug: Dapagliflozin — dapagliflozin tablet 2.5 mg Oral Single dose
  Arms: 1; 2
Drug: Metformin — metformin IR tablet 850 mg Oral Single dose
  Other Names: Glucophage
  Arms: 1; 2
Drug: Dapagliflozin/Metformin — Fixed dose combination dapagliflozin/metformin IR tablet 5 mg/1000 mg Oral Single dose
  Arms: 3; 4
Drug: Dapagliflozin — dapagliflozin tablet 5 mg Oral Single dose
  Arms: 3; 4
Drug: Metformin — metformin IR tablet 1000 mg Oral Single dose
  Other Names: Glucophage
  Arms: 3; 4

SUMMARY:
The primary objective of the study is to establish if the same amount of drug is absorbed into the blood after ingesting a combination dapagliflozin/metformin tablet vs. the individual dapagliflozin tablet and individual metformin tablet.

ELIGIBILITY:
Inclusion Criteria:

* Female healthy volunteers must be post-menopausal (cessation of menses >1year), be surgically sterile (documented) or hysterectomy or on abstinence
* Have normal physical exam, vital signs Electrocardiogram (ECG) findings, and laboratory values

Exclusion Criteria:

* Use of prescription medication for a chronic or acute medical condition within 3 weeks of randomization
* History of allergy to metformin
* Previous participation in an AstraZeneca (AZ) or BristolMyers-Sqibb dapagliflozin study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
bioequivalence will be demonstrated if the 90% confidence interval (CI) for the formulation effect is contained within the interval of 0.8000-1.2500 for AUC(0-t), AUCinf and Cmax with respect to both dapagliflozin and metformin. | Immediately prior to administration of the investigational product (IP). After intake of IP PK blood samples will be drawn every 15 minutes for the first hour, every 30 minutes for the second hour and every hour up to 72 h after intake of IP.

SECONDARY OUTCOMES:
To examine the safety and tolerability of the combination of dapagliflozin and metformin. | Throughout study (for 4 days in each period and a follow-up visit ~6 days later)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Golor, M.D., Principal Investigator — Parexel; Thomas Koernicke, Study Director — Parexel
Locations (1):
- Research Site, Berlin, Germany